CLINICAL TRIAL: NCT02218944
Title: Response Inhibition Training in Smoking Cessation
Brief Title: Smoking Response Inhibition Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: North Dakota State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SM14171
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Response Inhibition Training: A (Experimental): In the experimental condition, 20% of responses are no-go, with the majority of no-go responses paired with smoking images.
  Interventions: Behavioral: Response Inhibition Training
- Response Inhibition Training: B (Active Comparator): In the active comparator condition, 20% of responses are no-go trials, with no-go responses spread evenly across the various images.
  Interventions: Behavioral: Response Inhibition Training
- Benign (Placebo Comparator): A benign condition has also been added to control for the possibility that response inhibition training, regardless of target, increases behavioral control and hence decreases relapse likelihood. The benign condition has 50% no-go trials, with no-go responses spread evenly across images.

INTERVENTIONS:
Behavioral: Response Inhibition Training — The primary purpose of this research is to examine the feasibility and efficacy of a smoking specific response inhibition training program in the context of a quit attempt. The task is based on a modified stop-signal task. The study utilizes a one-way nested design with three conditions.
  Other Names: Stop-signal Task; Go/No-Go Task
  Arms: Response Inhibition Training: A; Response Inhibition Training: B

SUMMARY:
The current study tests a response inhibition retraining program, implemented on a mobile device, as a mechanism to increase relapse prevention during a smoking cessation attempt. Study participants (n = 150) are randomly assigned to a control, benign, or intervention condition. They complete 2 weeks of response inhibition retraining, and then engage in a cessation attempt. It is hypothesized that individuals who receive the intervention will have a decreased likelihood of relapse following the cessation attempt. In addition, it is hypothesized that this is due to decreases in implicit smoking motivation as a function of the response inhibition training.

DETAILED DESCRIPTION:
Smoking is the leading preventable cause of death and disease in the U.S. Each year approximately 30% of smokers try to quit, with the vast majority of attempts (~90%) ending in relapse. This is complicated by treatment barriers related to cost and accessibility. Identifying cost effective ways to aide in cessation success, which can be widely disseminated, remains vitally important. According to the dual-process model of substance use, addiction develops via an imbalance between effortful control and automatic psychological processes. The affective processing model suggests that during withdrawal, automatic psychological processes increase implicit drug seeking motivation. Implicit motivation is hypothesized as the underlying mechanism through which automatic psychological processes exert control over behavior. Research suggests that behavioral impulse control may attenuate the association between implicit motivation and substance use. Response inhibition, one form of behavioral impulse control, is the ability to inhibit behavioral responses to salient approach cues. Smokers tend to have less behavioral impulse control. In addition, poor behavioral impulse control makes individuals more vulnerable to various risk factors associated with relapse (e.g., positive expectancies, higher craving during abstinence, etc.). Improving smoking relevant behavioral impulse control may affect multiple indices of relapse. Research in cognitive retraining has shown that response inhibition can be modified through training. Recently this has been extended to training using mobile devices. The development of mobile interventions which specifically target underlying mechanisms of addiction may provide a novel adjunct to current cessation programs. The current proposal builds on previous research by implementing a response inhibition training paradigm in the context of a cessation trial. It is hypothesized that this task will reduce the likelihood of relapse following a quit attempt. Furthermore, it is hypothesized that training effects will operate via decreases in implicit motivation and global craving. If successful, the current study will provide evidence for a relapse prevention tool that can (1) increase overall cessation success and (2) be widely and easily dispersed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18-45 years old, who smoke at least 10 cigarettes/day, score 5 or higher on the Fägerstrom Test of Nicotine Dependence, express a desire to quit, and have no current psychiatric diagnoses.

Exclusion Criteria:

* Individuals will be ineligible to participate if they have used other tobacco products (e.g., smokeless tobacco) on more than 5 days in the past month, intend to quit smoking using pharmacotherapy, or are non-English speaking.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Smoking relapse | 6 months
  A relapse is defined as a resumption of smoking behavior, following a cessation attempt, with the acknowledgement that the study participant is no longer trying to quit smoking. Abstinence is verified with Cotinine.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Dvorak, PhD, Principal Investigator — Amy Scott, PhD
Locations (1):
- North Dakota State University, Fargo, North Dakota, United States